CLINICAL TRIAL: NCT03493919
Title: A Sourcing Study to Collect Human Biological (Serum) Samples From Healthy Adults
Brief Title: A Sourcing Study to Collect Human Blood Samples From Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 207911; 2017-002919-33 (EudraCT Number)
Record Dates: First submitted 2018-02-06; First posted 2018-04-11 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Meningitis, Meningococcal
Keywords: Immunological assays; Human blood donors; Meningococcal vaccination; Meningococcal disease
MeSH Terms: conditions — Meningitis, Meningococcal; Meningococcal Infections | interventions — 4CMenB vaccine; MenACWY; Meningococcal Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- rMenB+OMV NZ Group (Experimental): Participants vaccinated intramuscularly with Bexsero vaccine at Day 1 and Day 61 and blood samples were collected at Day -83, Day 8, and Day 98.
  Interventions: Biological: rMenB+OMV NZ vaccine
- MenACWY 1 Group (Experimental): Participants vaccinated intramuscularly with Menveo vaccine at Day 1 and blood samples were collected at Day -83, Day 8, and Day 151.
  Interventions: Biological: Meningococcal Groups A, C, W and Y Conjugate Vaccine (MenACWY)
- MenACWY 2 Group (Experimental): Participants vaccinated intramuscularly with Menveo vaccine at Day 1 and blood samples were collected at Day -60, Day 31, and Day 151.
  Interventions: Biological: Meningococcal Groups A, C, W and Y Conjugate Vaccine (MenACWY)
- MenACWY 3 Group (Experimental): Participants vaccinated intramuscularly with Menveo vaccine at Day 1 and blood samples were collected at Day -30, Day 61, and Day 151.
  Interventions: Biological: Meningococcal Groups A, C, W and Y Conjugate Vaccine (MenACWY)

INTERVENTIONS:
Biological: rMenB+OMV NZ vaccine — Two doses of rMenB+OMV NZ vaccine were administered intramuscularly at Day 1 and Day 61.
  Other Names: Bexsero
  Arms: rMenB+OMV NZ Group
Biological: Meningococcal Groups A, C, W and Y Conjugate Vaccine (MenACWY) — One dose of MenACWY vaccine were administered intramuscularly at Day 1.
  Other Names: Menveo
  Arms: MenACWY 1 Group; MenACWY 2 Group; MenACWY 3 Group

SUMMARY:
The purpose of this study was to collect large volumes of matched pairs of pre- and post-vaccination sera from healthy subjects who administered GlaxoSmithKline (GSK) Biologicals' vaccine against meningitis- MenACWY vaccine (Menveo) or rMenB+OMV NZ vaccine (Bexsero), which serves for the development, qualification, validation, and maintenance of immunological assays which supports the preclinical research activities and clinical development of GSK Biologicals' vaccines. The safety of the subjects given one of the two vaccines (Bexsero or Menveo), as per the recommended dosage and schedule were assessed during their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* A male or female between, and including, 18 and 50 years of age at the time of the first study visit.
* Healthy subjects as established by medical history and clinical examination before entering into the study. Healthy subjects with no medical conditions that, in the opinion of the investigator, prevents the subject from participating in the study.
* Subjects must weigh at least 110 pounds (50 kg), but not to present obesity (BMI < 32kg/m2).
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination and
  * has agreed to continue adequate contraception during the entire treatment period and for 1 month, after completion of the vaccination series.

Exclusion Criteria:

* Progressive, unstable or uncontrolled clinical conditions.
* Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Abnormal function of the immune system resulting from:

  * Clinical conditions.
  * Systemic administration of corticosteroids (PO/IV/IM) within 90 days prior to informed consent.
  * Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
* Received immunoglobulins or any blood products within 180 days prior to informed consent.
* Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.
* Any history of meningococcal vaccination or meningococcal and gonorrhoea diseases.
* Enrolment in any activity requiring a blood donation greater than 50 mL during the period starting 30 days before the first study visit (Day -83, Day -60 or Day -30) or for the duration of the study period.
* Administration of long-acting immune-modifying drugs at any time during the study period
* Subjects with blood disorders.
* Subjects with a history of difficulty in providing blood samples
* Any antibiotic intake 7 days prior to blood collection.
* Subjects who donated >450 mL of blood within 60 days prior to any blood collection visits.
* Subjects who lost >200 mL during a single apheresis or who lost red blood cells on more than one occasion during apheresis within the previous 60 days.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product
* Ongoing anaemia as indicated by haemoglobin values below the lower limit of the laboratory-specified reference range. If the finger prick method demonstrates an anaemia, no further protocol procedures will be performed, and the subject will be referred for appropriate medical management. The subject may participate in this study following therapy and evidence that the anaemia has been resolved.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition based on medical history and physical examination
* Family history of congenital or hereditary immunodeficiency.
* Serious chronic illness.
* History of chronic alcohol consumption and/or drug abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1021 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Australia (5):
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Spearwood, Western Australia
- GSK Investigational Site, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To comply with the local health authorities and guidelines [Australian Red Cross, 2016] with a minimum 90-day interval between blood draws, 3 MenACWY groups were formed to ensure blood draw at Days -83 [83 days before first vaccination (Day 1)], -60 [60 days before first vaccination (Day 1), -30 [30 days before first vaccination (Day 1), 31, 61, and 151. The rMenB+OMV NZ group was not split due to sufficient intervals between the post-vaccination blood sampling time points (Day 8 and Day 98).
Pre-assignment Details: Out of 1021 participants enrolled, 60 participants did not receive vaccination as they did not meet the eligibility criteria or withdrew from the study, therefore only 961 participants were included in the Exposed Set and started the study.
Period: Overall Study
Arm/Group | rMenB+OMV NZ Group | MenACWY 1 Group | MenACWY 2 Group | MenACWY 3 Group
Started | 470 | 165 | 165 | 161
Completed | 454 | 161 | 163 | 157
Not Completed | 16 | 4 | 2 | 4
Not completed — Other | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 9 | 3 | 1 | 1
Not completed — Lost to Follow-up | 5 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rMenB+OMV NZ Group | MenACWY 1 Group | MenACWY 2 Group | MenACWY 3 Group | Total
Number analyzed (Participants) | 470 | 165 | 165 | 161 | 961
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 32.8 (8.8) | 33.3 (9.1) | 33.3 (9.0) | 32.9 (8.8) | 33.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295 | 99 | 105 | 109 | 608
  Male | 175 | 66 | 60 | 52 | 353
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 29 | 13 | 15 | 8 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 430 | 150 | 149 | 147 | 876
  More than one race | 9 | 2 | 1 | 6 | 18
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Human Blood Samples Collected for Conversion Into Serum at Day -83
Description: The Serum Bactericidal Assay (SBA) using human serum used to measure the induction of functional bactericidal antibodies directed against Neisseria meningitidis. To comply with local health authorities and guidelines [Australian Red Cross, 2016], blood samples were collected with the minimum interval of approximately 90 days. For Day -83, blood samples were collected only for rMenB+OMV NZ group and MenACWY 1 group.
Time Frame: At Day -83 [83 days before first vaccination (Day 1)]
Population: Analysis was performed on blood samples collected from exposed set, which included all participants in the enrolled set who received a study vaccination. The participants included in this outcome measure are based on the data collected at specific blood sampling timepoints.
Measure: Number; unit: Blood samples
Units Other Than Participants: Samples
Arm/Group | rMenB+OMV NZ Group | MenACWY 1 Group
Number analyzed (Participants) | 470 | 165
Number analyzed (Samples) | 5578 | 1936
Blood samples | 5578 | 1936

2. Primary Outcome: Number of Human Blood Samples Collected for Conversion Into Serum at Day 8
Description: The Serum Bactericidal Assay (SBA) using human serum used to measure the induction of functional bactericidal antibodies directed against Neisseria meningitidis. To comply with local health authorities and guidelines [Australian Red Cross, 2016], blood samples were collected with the minimum interval of approximately 90 days. For Day 8, blood samples were collected only for rMenB+OMV NZ group and MenACWY 1 group.
Time Frame: At Day 8
Population: as for outcome 1
Measure: Number; unit: Blood samples
Units Other Than Participants: Samples
Arm/Group | rMenB+OMV NZ Group | MenACWY 1 Group
Number analyzed (Participants) | 462 | 162
Number analyzed (Samples) | 5396 | 1907
Blood samples | 5396 | 1907

3. Primary Outcome: Number of Human Blood Samples Collected for Conversion Into Serum at Day 98
Description: The Serum Bactericidal Assay (SBA) using human serum used to measure the induction of functional bactericidal antibodies directed against Neisseria meningitidis. To comply with local health authorities and guidelines [Australian Red Cross, 2016], blood samples were collected with the minimum interval of approximately 90 days. For Day 98, blood samples were collected only for rMenB+OMV NZ group.
Time Frame: At Day 98
Population: as for outcome 1
Measure: Number; unit: Blood samples
Units Other Than Participants: Samples
Arm/Group | rMenB+OMV NZ Group
Number analyzed (Participants) | 454
Number analyzed (Samples) | 5204
Blood samples | 5204

4. Primary Outcome: Number of Human Blood Samples Collected for Conversion Into Serum at Day 151
Description: The Serum Bactericidal Assay (SBA) using human serum used to measure the induction of functional bactericidal antibodies directed against Neisseria meningitidis. To comply with local health authorities and guidelines [Australian Red Cross, 2016], blood samples were collected with the minimum interval of approximately 90 days. For Day 151, blood samples were collected only for MenACWY 1, 2 and 3 group.
Time Frame: At Day 151
Population: as for outcome 1
Measure: Number; unit: Blood samples
Units Other Than Participants: Samples
Arm/Group | MenACWY 1 Group | MenACWY 2 Group | MenACWY 3 Group
Number analyzed (Participants) | 161 | 162 | 156
Number analyzed (Samples) | 1869 | 1866 | 1752
Blood samples | 1869 | 1866 | 1752

5. Primary Outcome: Number of Human Blood Samples Collected for Conversion Into Serum at Day -60
Description: The Serum Bactericidal Assay (SBA) using human serum used to measure the induction of functional bactericidal antibodies directed against Neisseria meningitidis. To comply with local health authorities and guidelines [Australian Red Cross, 2016], blood samples were collected with the minimum interval of approximately 90 days. For Day -60, blood samples were collected only for MenACWY 2 group.
Time Frame: At Day -60 [60 days before first vaccination (Day 1)]
Population: as for outcome 1
Measure: Number; unit: Blood samples
Units Other Than Participants: Samples
Arm/Group | MenACWY 2 Group
Number analyzed (Participants) | 165
Number analyzed (Samples) | 1957
Blood samples | 1957

6. Primary Outcome: Number of Human Blood Samples Collected for Conversion Into Serum at Day 31
Description: The Serum Bactericidal Assay (SBA) using human serum used to measure the induction of functional bactericidal antibodies directed against Neisseria meningitidis. To comply with local health authorities and guidelines [Australian Red Cross, 2016], blood samples were collected with the minimum interval of approximately 90 days. For Day 31, blood samples were collected only for MenACWY 2 group.
Time Frame: At Day 31
Population: as for outcome 1
Measure: Number; unit: Blood samples
Units Other Than Participants: Samples
Arm/Group | MenACWY 2 Group
Number analyzed (Participants) | 163
Number analyzed (Samples) | 1920
Blood samples | 1920

7. Primary Outcome: Number of Human Blood Samples Collected for Conversion Into Serum at Day-30
Description: The Serum Bactericidal Assay (SBA) using human serum used to measure the induction of functional bactericidal antibodies directed against Neisseria meningitidis. To comply with local health authorities and guidelines [Australian Red Cross, 2016], blood samples were collected with the minimum interval of approximately 90 days. For Day -30, blood samples were collected only for MenACWY 3 group.
Time Frame: At Day -30 [30 days before first vaccination (Day 1)]
Population: as for outcome 1
Measure: Number; unit: Blood samples
Units Other Than Participants: Samples
Arm/Group | MenACWY 3 Group
Number analyzed (Participants) | 161
Number analyzed (Samples) | 1894
Blood samples | 1894

8. Primary Outcome: Number of Human Blood Samples Collected for Conversion Into Serum at Day 61
Description: The Serum Bactericidal Assay (SBA) using human serum used to measure the induction of functional bactericidal antibodies directed against Neisseria meningitidis. To comply with local health authorities and guidelines [Australian Red Cross, 2016], blood samples were collected with the minimum interval of approximately 90 days. For Day 61, blood samples were collected only for MenACWY 3 group.
Time Frame: At Day 61
Population: as for outcome 1
Measure: Number; unit: Blood samples
Units Other Than Participants: Samples
Arm/Group | MenACWY 3 Group
Number analyzed (Participants) | 159
Number analyzed (Samples) | 1809
Blood samples | 1809

9. Secondary Outcome: Number of Participants With Atleast One Serious Adverse Events (SAEs) Related to Vaccination
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of hospitalization, results in disability/incapacity in a subject or is a congenital anomaly/ birth defect in the offspring of a study subject. AE(s) considered as SAE(s) also include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, as per the medical or scientific judgement of the physician. Related=AE assessed by the investigator as related to the vaccination.
Time Frame: Throughout the study period (approximately 4 years)
Population: Analysis was performed on blood samples collected from exposed set, which included all participants subjects in the exposed set who provide safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | rMenB+OMV NZ Group | MenACWY 1 Group | MenACWY 2 Group | MenACWY 3 Group
Number analyzed (Participants) | 470 | 165 | 165 | 161
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were collected throughout the study period (Up to 4 years)
Description: According to the pre-specified protocol, only serious adverse events and pregnancy-related events were to be collected. As no pregnancies have been reported in this study, the total number of participants at risk and affected by any other adverse events is zero.
Arm/Group | rMenB+OMV NZ Group | MenACWY 1 Group | MenACWY 2 Group | MenACWY 3 Group
All-Cause Mortality (participants affected / at risk) | 0/470 | 0/165 | 0/165 | 0/161
Serious Adverse Events (participants affected / at risk) | 3/470 | 1/165 | 1/165 | 0/161
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rMenB+OMV NZ Group (N=470) | MenACWY 1 Group (N=165) | MenACWY 2 Group (N=165) | MenACWY 3 Group (N=161)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03493919/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03493919/SAP_001.pdf